CLINICAL TRIAL: NCT00648492
Title: Single-Dose Food In Vivo Bioequivalence Study Metformin Hydrochloride ER Tablets (500 mg; Mylan) and Glucophage® XR (500 mg; Bristol-Myers Squibb) in Healthy Volunteers
Brief Title: Food Study Metformin Hydrochloride ER Tablets 500 mg and Glucophage® XR 500 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: METF-0284
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin

ARMS (2):
- 1 (Experimental): Metformin Hydrochloride ER Tablets 500 mg
  Interventions: Drug: Metformin Hydrochloride ER Tablets 500 mg
- 2 (Active Comparator): Glucophage® XR 500 mg
  Interventions: Drug: Glucophage® XR 500 mg

INTERVENTIONS:
Drug: Metformin Hydrochloride ER Tablets 500 mg — 500mg, single dose fed
  Arms: 1
Drug: Glucophage® XR 500 mg — 500mg, single dose fed
  Arms: 2

SUMMARY:
The objective of this study is to investigate the bioequivalence of Mylan's metformin hydrochloride ER tablets to Bristol-Myers Squibb's Glucophage® XR tablets following a single, oral 500 mg (1 x 500 mg) dose administered under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older.
2. Sex: Male and non-pregnant, non-lactating female

   1. Women of childbearing potential must have negative serum (Beta HCG) pregnancy tests performed within 14 days prior to the start of the study and on the evening prior to each dose administration. If dosing is scheduled on Sunday or Monday, the HCG pregnancy test should be given within 48 hours prior to dosing of each study period. An additional serum (Beta HCG) pregnancy test will be performed upon completion of the study.
   2. Women of childbearing potential must practice abstinence or be using an acceptable form of contraception throughout the duration of the study. Acceptable forms of contraception include the following:

      1. intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or
      2. barrier methods containing or used in conjunction with a spermicidal agent, or
      3. postmenopausal accompanied with a documented postmenopausal course of at least one year or surgical sterility (tubal ligation, oophorectomy or hysterectomy).
   3. During the course of the study, from study screen until study exit - including the washout period, women of childbearing potential must use a spermicide containing barrier method of contraception in addition to their current contraceptive device. This advice should be documented in the informed consent form.
3. Weight: At least 60 kg (132 lbs) for man and 48 kg (106 lbs) for women and within 15% of Ideal Body Weight (IBW), as referenced by the Table of ""Desirable Weights of Adults"" Metropolitan Life Insurance Company, 1999 (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
4. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, laboratory evaluation, 12-lead ECG, hepatitis B and hepatitis C tests, HIV test, and urine drug screen including amphetamine, barbiturates, benzodiazepine, cannabinoid, cocaine, opiates, phencyclidine, and methadone) performed within 14 days of the initial dose of study medication.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco products.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within the 48 hours prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. Positive test for any drug included in the urine drug screen.
3. Medications:

   1. Use of any medication within the 14 days prior to the initial dose of study medication.
   2. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
   3. Use of hormonal contraceptives and hormonal replacement therapy within three months prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant chronic disease and/or hepatitis.
   2. History of drug and/or alcohol abuse.
   3. Acute illness at the time of either the prestudy medical evaluation or dosing.
   4. Positive HIV, Hepatitis B, or Hepatitis C test.
   5. Renal disease or renal dysfunction (as suggested by serum creatinine levels greater than or equal to 1.5 mg/dL (for males) and greater than or equal to 1.4 mg/dL (for females) or abnormal creatinine clearance).
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide for Clinically Relevant Abnormalities (see Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to metformin hydrochloride.
9. History of difficulty in swallowing medication, or any gastrointestinal disorder which could affect the drug absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-10; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D., Principal Investigator — PRACS Institute Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html